CLINICAL TRIAL: NCT05848479
Title: Effect of Clamshell Exercise on Lumbopelvic Stability and Low Back Pain in Post Partum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eman Mahmoud Mahmoud El-sayed Ellily (Other)
Responsible Party: Sponsor-Investigator, Eman Mahmoud Mahmoud El-sayed Ellily, post graduate researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004341
Record Dates: First submitted 2023-04-06; First posted 2023-05-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lumbosacral Instability; Low Back Pain Post Partum
Keywords: clamshell exercise; lumbopelvic instability; low back pain; post partum
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Abdominal bracing
  Interventions: Other: Abdominal bracing
- study group (Active Comparator): Abdominal bracing and clamshell exercise
  Interventions: Other: Abdominal bracing; Other: clamshell exercise

INTERVENTIONS:
Other: Abdominal bracing — they will perform 3 times/week of static abdominal contraction for six weeks.
Other: clamshell exercise — Each women will be positioned in side lying on the floor, with the pelvis and the spine in neutral position, the hips will bent at 45° and the knees flexed to 90°. She will abduct the top knee as far as possible, while keeping the heels together, then return to the starting position , the position will be maintained for 5 seconds in an abduction state, and repeated 10 times, with rest for 1 minute to minimize muscle fatigue,they will perform 3 times/week fo 6 weeks
  Arms: study group

SUMMARY:
This study will be conducted on 44 females with postpartum LBP & pelvic instability, selected from Dar of women hospital in port said to investigate effect of clamshell exercise on lumbo-pelvic stability and low back pain in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

1. Post-partum females complaining of LBP and lumber instability
2. Their age will be ranged from 25-35 years.
3. Their BMI will be ranged from 25-30 kg/m2

Exclusion Criteria:

1. Spinal deformity.
2. Lower limb deformity.
3. Osteosarcoma
4. Mental disorders. 5-25>BMI>30

6-Performing any physical exercise at the time of the study. 7-Bad general Health

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2023-05-26 (Estimated); Primary Completion 2023-07-26 (Estimated); Study Completion 2023-07-26 (Estimated)

PRIMARY OUTCOMES:
Change in the degree of lumbopelvic instability | change in the lumbopelvic instability degree will be measured at baseline and after 6 weeks of the interventions
  Change in the degree of lumbopelvic instability will be measured by specific tests(The dip test, the runner pose test and the single leg squat test) and the pateint performance will be graded as poor or good
lumbopelvic range of motion | change in the lumbopelvic instability degree will be measured at baseline and after 6 weeks of the interventions
  Degree of lumbopelvic range of motion will be measured by goniometer

SECONDARY OUTCOMES:
severity of pain intensity | change in the lumbopelvic instability will be measured at baseline and after 6 weeks of the interventions
  change in low back pain intensity will be measured using visual analogue scale(VAS)
  low back pain intensity
the degree of function disability | change in the lumbopelvic instability will be measured at baseline and after 6 weeks of the interventions
  the change in the degree of function disability will be measured by Oswestry disability index (ODI)

IPD SHARING:
Plan to Share IPD: No